CLINICAL TRIAL: NCT01050790
Title: Lenalidomide and Azacitidine for Adaptive Immunotherapy in Multiple Myeloma: Pilot Study of Autologous Lymphocyte Mobilization Following Immuno-modulatory Therapy
Brief Title: Lenalidomide + Azacitidine for Adaptive Immunotherapy -> Auto SCT in Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000663409; P30CA016059 (NIH); MCC-12430 (Other: Massey Cancer Center)
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2016-10

CONDITIONS: Multiple Myeloma
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aza Len Lymphapheresis SCT ALI (Experimental): Azacitidine will be administered to all the patients subcutaneously at a dose of 75 mg/m2 daily for five days(day 1-5). These cycles will be repeated at 28 day intervals depending on hematopoietic recovery. Starting on day 6 patients will receive lenalidomide 15 mg PO daily until day 21. No drug will be administered from day 22 to day 28. Lymphapheresis will occur after cycles 2 and 3.Patients will undergo a stem cell collection approximately two weeks after complete myeloid recovery from the third cycle of therapy. Stem Cell Transplant (SCT) will occur per transplant center protocols. Post-transplant single or tandem autologous lymphocyte infusions (ALI) will be performed no earlier than 30 days post-transplant and no later than 40 days.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Subject will receive Vidaza (azacitidine) and Revlimid (lenalidomide) as treatment for their multiple myeloma. The Vidaza will be given for 5 days as an injection. On day 6 they will receive Revlimid taken by mouth every day for 16 days followed by 7 days of rest. The drug cycle will be repeated 0, 1 or 2 more times depending on how their blood counts recover.
  Other Names: Vidaza®; lenalidomide; CC-5013; Revlimid

SUMMARY:
RATIONALE: Lenalidomide may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. An autologous stem cell transplant may be able to replace blood-forming cells that were destroyed by lenalidomide and azacitidine. Giving autologous lymphocytes after the transplant may help destroy any remaining cancer cells.

PURPOSE: This pilot trial is studying how well giving lenalidomide together with azacitidine works when followed by autologous stem cell transplant and autologous lymphocyte infusion in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of mobilizing and infusing autologous lymphocytes (ALI) following immunomodulatory therapy comprising azacitidine and lenalidomide in patients with multiple myeloma.

Secondary

* Determine the ability to proceed with autologous stem cell transplantation in these patients.
* Determine the complete response rate at 6 months following transplant in patients treated with this regimen.
* Determine the progression-free survival and overall survival of patients treated with this regimen.
* Determine the time to progression in patients treated with this regimen.
* Monitor the toxicity of post-autologous stem cell infusion of autologous lymphocytes.
* Measure the pre- and post-ALI immune response to cancer testis antigens (CTA) (CTA-specific Ig and T-cell repertoire).
* Study the expression of CTA in multiple myeloma before and after azacitidine therapy.

OUTLINE:

* Immunomodulatory therapy: Patients receive azacitidine subcutaneously on days 1-5 and oral lenalidomide on days 6-21. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
* Lymphapheresis: Patients undergo autologous lymphocyte harvest on day 22 of courses 2 and 3.
* Autologous stem cell transplantation (ASCT): Patients undergo single or tandem ASCT using standard protocols.
* Autologous lymphocyte infusion (ALI): Patients undergo ALI approximately 28-60 days after ASCT.

Blood samples are collected at baseline and periodically during study for correlative laboratory studies, including CTA-specific immune monitoring by RT-PCR, ELISPOT assays, and flow cytometry. Tissue samples from bone marrow aspirates are also collected at baseline, during course one, and after course three for CTA expression and methylation studies.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Inclusion criteria:

* Patients with a diagnosis of multiple myeloma, who have residual measurable disease (in partial remission or with stable disease) and are eligible to undergo an autologous stem cell transplant will be able to participate in this trial; measurable disease will comprise of either, quantifiable serum or urinary, M protein or free light chains in the presence of a positive immunofixation or bone marrow plasma cells > 5%
* Patients who have received prior lenalidomide therapy will be eligible if >= partial response (PR) was observed on a prior lenalidomide containing regimen and patients did not progress while receiving lenalidomide; isolated bone lytic lesions in the absence of measurable para-proteins will not be considered measurable disease
* A minimum period of two weeks must have elapsed following the prior myeloma therapy; this does not include therapy with bisphosphonates
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* No clinical evidence of uncontrolled viral, fungal, bacterial infection
* Negative serology for human immunodeficiency virus (HIV)
* Serum bilirubin =< 1.5 times upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT)/serum glutamic pyruvic transaminase (SGPT) =< 3x ULN
* Calculated creatinine clearance >= 60ml/min by Cockcroft-Gault formula; creatinine clearance >= 60 ml/min or serum creatinine =< 2.0 mg/dL
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelet count >= 100,000/ uL
* Hemoglobin (Hgb) >= 10 g/dL following recovery from last therapy
* Cardiac and pulmonary function adequate for transplant
* Ability to sign informed consent
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy

Exclusion criteria:

* Known or suspected hypersensitivity to azacitidine or mannitol
* Patients with multiple myeloma refractory to therapy with lenalidomide; progression following discontinuation of prior therapy with lenalidomide is allowed as long as patients have not failed rechallenge with lenalidomide
* Pregnant or breast feeding
* Other concomitant malignancies
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Concurrent use of other anti-cancer agents or treatments
* Known hypersensitivity to thalidomide or lenalidomide

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-01; Primary Completion 2014-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir A. Toor, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Result] Toor AA, Payne KK, Chung HM, Sabo RT, Hazlett AF, Kmieciak M, Sanford K, Williams DC, Clark WB, Roberts CH, McCarty JM, Manjili MH. Epigenetic induction of adaptive immune response in multiple myeloma: sequential azacitidine and lenalidomide generate cancer testis antigen-specific cellular immunity. Br J Haematol. 2012 Sep;158(6):700-11. doi: 10.1111/j.1365-2141.2012.09225.x. Epub 2012 Jul 23. PMID 22816680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential patients will be identified at the first BMT consult. They will then be preliminarily screened. If deemed eligible, they will be consented at the second BMT consult. After consent the subject will be officially screened for eligibility as described in the protocol. If eligible they will be enrolled.
Period: Overall Study
Arm/Group | Aza Len Lymphapheresis SCT ALI
Started | 17
Completed | 16
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Multiple Myeloma in either first or subsequent partial remission with measurable disease, eligible for autologous SCT.
Arm/Group | Aza Len Lymphapheresis SCT ALI
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.59 (7.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Feasibility to Mobilize and Infuse Autologous Lymphocytes (ALI) After Immunomodulatory Therapy and After Stem Cell Transplant Engraftment
Description: Time frame is post 2nd and 3rd cycles of rev/aza and after stem cell transplant engraftment.
Time Frame: 6 months
Population: 17 of 17 patients were able to mobilize lymphocytes. 16 of 17 patients had lymphocytes infused post transplant. 1 patient was not able to mobilize stem cells and so did not go to transplant.
Measure: Number; unit: participants
Groups:
- 5-azacytidine + Lenalidomide -> Auto Stem Cell Transplant: azacitidine: 75 mg/sq m daily for 5 days
  lenalidomide: 10 mg p.o. daily, Days 6-21
Arm/Group | 5-azacytidine + Lenalidomide -> Auto Stem Cell Transplant
Number analyzed (Participants) | 17
participants
  mobilize lymphocytes | 17
  lymphocytes infused post transplant | 16
  not able to mobilize stem cells/no transplant | 1

2. Secondary Outcome: Complete Response Rate at 6 Months
Description: 16 of 17 patients proceeded to transplant. 6 month CR rate post transplant was 8/16 (50%).
Time Frame: 6 months
Population: 1 patient did not proceed to transplant.
Measure: Number; unit: percentage of participants
Arm/Group | 5-azacytidine + Lenalidomide -> Auto Stem Cell Transplant
Number analyzed (Participants) | 16
percentage of participants | 50

3. Secondary Outcome: Toxicity as Assessed by NCI CTCAE v3.0
Description: Time frame includes after stem cell transplant engraftment. Toxicity post ALI infusion: 1 patient grade 1 hypertension 90 min post infusion. Toxicity post Rev maintenance: 1 patient not tolerated, 1 patient dose decreased due to counts.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | 5-azacytidine + Lenalidomide -> Auto Stem Cell Transplant
Number analyzed (Participants) | 17
participants
  Toxicity post ALI infusion | 1
  Toxicity post Rev maintenance | 2

4. Secondary Outcome: Time to Progression Post Transplant
Description: Time to progression post transplant: For patients not in Complete Response (CR), progressive disease requires one or more: >25% increase in the level of the serum monoclonal paraprotein(absolute increase of at least 0.5 g/dL); > 25% increase in 24-hour urinary light chain excretion(absolute increase of at least 200m/24 hours). Increase plasma cells in a bone marrow aspirate( absolute increase of at least 10%). Definite increase in the size of existing bone lesions or soft tissue plasmacytomas. Development of new bone lesions or soft tissue plasmacytomas. Development of hypercalcemia (corrected serum Ca > 11.5 mg/dL or > 2.65 mmol/L) not attributable to any other cause. All relapse categories require two consecutive assessments made any time before classification as relapse or progressive disease.
Time Frame: 28 months
Population: Progression is collected anytime after transplant.
Measure: Median (Full Range); unit: months
Arm/Group | 5-azacytidine + Lenalidomide -> Auto Stem Cell Transplant
Number analyzed (Participants) | 17
months | 14.9 [4.2 to 28.1]

5. Secondary Outcome: Progression-free and Overall Survival
Description: Survival and event-free survival curves (any event of fatality, relapse, acute or chronic GVHD) with Kaplan-Meier curves. The incidence curve for relapse - accounting for the competing risk of fatality - is plotted with step-wise curves. The R statistical software (version 2.15) was used for all time-to-event analyses, with the survival package used for survival curves, and the cmprsk package used for all competing risk curves.
  Results: The one-year survival rate is 93.3% (SE = 0.4%), and the two-year survival rate is 86.1% (SE = 0.9%).
Time Frame: 1 year to 2 years
Population: The outcome measure data was collected up to one to two years post transplant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-azacytidine + Lenalidomide -> Auto Stem Cell Transplant
Number analyzed (Participants) | 17
percentage of participants
  one- year survival rate | 93.3 [92.52 to 94.08]
  two-year survival rate | 86.1 [84.34 to 87.86]
  one-year relapse rate | 12.5 [11.13 to 13.87]
  two-year relapse rate | 19.2 [17.04 to 21.36]
  one-year event free survival rate | 87.5 [86.13 to 88.87]
  two-year event free survival rate | 67.3 [64.16 to 70.44]

6. Secondary Outcome: Pre- and Post-ALI Immune Response to Cancer Testis Antigens (CTA)
Description: Not able to obtain outcome data.
Time Frame: 6 months
Population: Not able to obtain outcome data. The lab doing this correlative analysis lost the personnel support to process the samples.
Arm/Group | Aza Len Lymphapheresis SCT ALI
Number analyzed (Participants) | 0

7. Secondary Outcome: CTA Expression Before and After Azacitidine Therapy
Description: Six patients tested have demonstrated CTA up-regulation in either unfractionated bone marrow (n = 4) or CD138+ cells (n = 2). CTA (CTAG1B)-specific T cell response has been observed in all three patients tested and persists following SCT.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | 5-azacytidine + Lenalidomide -> Auto Stem Cell Transplant
Number analyzed (Participants) | 17
participants
  CTA up-regulation | 6
  CD138+ cells | 2
  unfractionated bone marrow | 4
  CTA (CTAG1B)-specific T cell response | 3

ADVERSE EVENTS:
Time Frame: 1 year the subject will be on study and evaluated for adverse events.
Description: Medical history and physical before treatment, Days 1, 5 and 22 of the 1st cycle and before cycles 2 and 3, before ALI. Blood for study specific tests drawn before ALI and 2, 4 and 8 weeks after and if relapse occurs. Chest x ray before ALI. Bone marrow Biopsy at baseline and after cycle 3.
Arm/Group | 5-azacytidine + Lenalidomide -> Auto Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 9/17
Other Adverse Events (participants affected / at risk) | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-azacytidine + Lenalidomide -> Auto Stem Cell Transplant (N=17)
Pain - Pack (Musculoskeletal and connective tissue disorders) | 1 (1) — Hospitalization. Received radiation therapy with improvement. Grade 3: Severe pain; pain or analgesics severely interfering with ADL.
Renal failure (Renal and urinary disorders) | 1 (1) — Hospitalization, disease progression and death occurred after 100 days. Grade 5, death.
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (1) — Hospitalization. Grade 3, Severe pain; pain or analgesics severely interfering with ADL.
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3, Symptomatic, interfering with ADL; O2 indicated.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Hospitalization.
Mood alteration - Anxiety (Psychiatric disorders) | 1 (1) — Neurology, Grade 2: Mild mood alteration not interfering with function .
Infection with normal ANC or Grade 1 or 2 neutrophils - blood (Blood and lymphatic system disorders) | 2 (2) — Hospitalization.
Hypotension (Cardiac disorders) | 1 (2) — Hospitalization.
Mental Status (Psychiatric disorders) | 1 (1) — Neurology. Hospitalization.
Hypertension (Cardiac disorders) | 1 (1) — Hospitalization. Grade 3: Requiring more than one drug or more intensive therapy than previously.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-azacytidine + Lenalidomide -> Auto Stem Cell Transplant (N=17)
Low Hemoglobin (Blood and lymphatic system disorders) | 2 (3) — Grade 2-3.
Neutropenia (Blood and lymphatic system disorders) | 11 (27) — Grade 2-3.
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4) — Grade 2-3.
High Creatinine (Blood and lymphatic system disorders) | 1 (4) — Grade 2-3.
High AST (Blood and lymphatic system disorders) | 1 (1) — Grade 2-3.
High ALT (Blood and lymphatic system disorders) | 1 (1) — Grade 2-3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes